CLINICAL TRIAL: NCT02499341
Title: Comparison Between Ketamine and Tramadol for Pain Management After Major Upper Abdominal Surgery
Brief Title: A Comparison Study Between Ketamine Versus Tramadol for Pain Management After Major Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Professor of Anesthesiology, MD, PhD, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 637
Record Dates: First submitted 2015-07-12; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain
Keywords: Tramadol; Ketamine; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Ketamine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Tramadol (Active Comparator): Intraoperative administration of a bolus dose of tramadol and continuous intravenous infusion of tramadol for up to 48 h postoperatively.
  Interventions: Drug: Tramadol
- Ketamine (Active Comparator): Intraoperative administration of a bolus dose of ketamine and continuous intravenous infusion of ketamine for up to 48 h postoperatively.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Tramadol — Tramadol administered intravenously (1mg/kg) thirty minutes before the expected end of surgery, followed by a continuous infusion of tramadol (0.2mg•kg-¹•h-¹) for up to 48 h after major upper abdominal surgery, in patients receiving PCA morphine postoperatively at a bolus dose of 1 mg with a lockout period of 8 minutes.
  Other Names: Tramal
  Arms: Tramadol
Drug: Ketamine — Ketamine administered intravenously (0.5mg/kg) thirty minutes before the expected end of surgery, followed by a continuous infusion of ketamine (0.12mg•kg-¹•h-¹) for up to 48 h after major upper abdominal surgery, in patients receiving PCA morphine postoperatively at a bolus dose of 1 mg with a lockout period of 8 minutes.
  Other Names: Ketalar
  Arms: Ketamine

SUMMARY:
The purpose of the study is the comparison between ketamine and tramadol, regarding the analgesia quality and efficiency, in patients receiving Patient Controlled Analgesia (PCA) morphine, after major upper abdominal surgeries such as hepatectomies, gastrectomies, Whipple procedures and peripheral pancreatectomies. The goal is to bring out an improved analgesia scheme, which can be applied to the clinical work and refine the analgesia provided for major procedures which require increased postoperative opioids doses. In the study, half of patients will receive continuous intravenous infusion of tramadol and Patient Controlled Analgesia morphine and the other half will receive continuous intravenous infusion of ketamine and Patient Controlled Analgesia morphine postoperatively after major upper abdominal surgery. The successful combination of different drugs targets at the improvement of the analgesia provided, the reduction of complications and the exploitation of the pharmacodynamic properties of each drug.

DETAILED DESCRIPTION:
This is a single blind, prospective, randomized controlled trial. Forty two adults patients of American Society of Anesthesiologists (ASA) physical status I-II, aged 18-70yr, scheduled for elective upper abdominal surgery under general anaesthesia are recruited. Signed informed consent is obtained from all patients. Patients are randomized into two groups.

1. Ketamine group: thirty minutes before the expected end of surgery, ketamine is administered IV at a load dose of 0.5mg/kg followed by a continuous infusion of ketamine (0.12mg•kg-¹•h-¹) for up to 48 h.
2. Tramadol group: thirty minutes before the expected end of surgery, tramadol is administered IV at a load dose of 1mg/kg followed by a continuous infusion of tramadol (0.2mg•kg-¹•h-¹) for up to 48 h.

The evening before the elective surgery, all patients are premedicated with 150 mg ranitidine and 100mg hydroxyzine orally and provided with instructions on how to use the PCA device. They are also explained the Visual Analogue Scale (VAS: 0-10).

All participants received the same protocol of general anaesthesia. Before the induction of anaesthesia all patients received metoclopramide 10 mg, ranitidine 50 mg and dimethindene 4 mg intravenously. Anaesthesia was induced with propofol 2 mg/kg, and fentanyl 2 mcg/kg, while the administration of rocuronium facilitates the trachea intubation. The anaesthesia maintenance is attained through continuous infusion of propofol 1%. After the induction of anaesthesia and before the surgical incision, patients receive 3 mcg/kg fentanyl and 0.1mg/kg morphine intravenously, while repetitive doses of morphine 0.05 mg/kg are administered in order to keep intraoperative systolic arterial pressure and heart rate within the range of 20% of the baseline values. The total morphine consumption is recorded.

Thirty minutes before the expected end of surgery, paracetamol 1gr is administered intravenously. Consequently, patients receive either ketamine or tramadol according to the study group, at the aforementioned bolus and continuous infusions doses. The pump remained attached to the intravenous line for 48 hours.

After the anaesthesia recovery patients are transferred to the Postanaesthesia Care Unit, where pain is assessed using the VAS (0-10) and treated with morphine bolus doses of 2 mg IV to achieve VAS scores <4. When VAS score <4 is attained, a PCA morphine pump is connected to a peripheral intravenous line and set to deliver morphine at a bolus dose of 1 mg with a lockout period of 8 minutes.

When patients are full recovered and stabilized, are transferred to the wards. Postoperative analgesia consisted of PCA morphine and continuous infusion of either ketamine in the ketamine-group or tramadol in the tramadol-group, respectively. If analgesia is not adequate and VAS >5, morphine rescue doses of 2 mg are given intravenously. If the repetitive morphine doses are not efficient, the interval time of the PCA morphine pump is set at 6 minutes. Metoclopramide 10 mg is prescribed to be given intravenously twice a day. Postoperative nausea and vomiting (PONV) is assessed with a 5-points scale (0-4). If PONV is >2, dexamethasone 8 mg is given as first line treatment, while ondansetron 4 mg is the second line treatment. Itching is treated with propofol 10 mg IV. If the symptom continues, the patient is removed from the study.

The study period is 48 hours (1, 2, 4, 6, 12, 18, 24, 36 and 48 hours) considering as zero time, the time of the connection of the PCA morphine pump to the patient. At these time points, morphine consumption, VAS scores, oxygen saturation, respiratory rate, bradycardia, hypotension, postoperative day of patient's mobilization, complications, drugs' side effects (itching, seizures, illusions, confusion, disorientation, sense of dry mouth, urinary retention, sedation, quality of sleep, PONV,) ability to cough are assessed. Additionally, patient's overall satisfaction at 48 hours is assessed and the postoperative total intrahospital stay is also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* American Society of Anesthesiologists (ASA) physical status I and II
* Major Upper abdominal Surgery (Elective Hepatectomy, Gastrectomy, Whipple procedure, Peripheral Pancreatectomy)

Exclusion Criteria:

* Patient's refusal to participate in the study
* Performance of regional anaesthesia
* Unsuitability for Patient Controlled Analgesia
* Current opiates use
* Drug addiction
* Chronic Pain Syndromes
* Alcohol addiction
* Epilepsy
* Psychiatric disorders
* Use of Monoamine Oxidase Inhibitor or Selective Serotonin Reuptake Inhibitor
* Sleep Apnea Syndrome
* Extrapyramidal Syndromes
* Severe liver, kidney or heart disease
* Known allergy to ketamine, tramadol or morphine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Measurement of morphine consumption expressed as milligrams postoperatively in abdominal surgery. | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Matsota, MD, PhD, Principal Investigator — Attikon University Hospital, Athens, Greece
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece